CLINICAL TRIAL: NCT02101567
Title: A Comparison Between Carbetocin, Oxytocin and Ergometrine in Prevention of Postpartum Haemorrhage Following Caesarean Section
Brief Title: Carbetocin Versus Oxytocin and Ergometrine for the Prevention of Postpartum Haemorrhage Following Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Lecturer of Obstetrics and Gynecology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Beni-Suef 3
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Bleeding; Anemia
Keywords: Postpartum hemorrhage, Cesarean section, Uterotonics
MeSH Terms: conditions — Hemorrhage; Anemia; Postpartum Hemorrhage | interventions — carbetocin; Oxytocin; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pabal ( carbetocin) (Active Comparator): Pabal (carbetocin which is a long acting oxytocin ) given as 100 mcg slow i.v. injection over 1 minute ( Draxis/Multiph). It will be given to the patients included in the study after delivery of the fetal head.
  Interventions: Drug: Pabal 100 mcg iv infusion over 1 minute given after delivery of fetal head
- Oxytocin and Methergine (methyl ergometrine) (Active Comparator): The second group of patients included in the study will be given Oxytocin 5 IU ampoule by intravenous infusion and Methergine 0.2 mg IV after delivery of fetal head.
  Interventions: Drug: Oxytocin 5 IU iv infusion and Methtergine 0.2 mg iv

INTERVENTIONS:
Drug: Pabal 100 mcg iv infusion over 1 minute given after delivery of fetal head — In the first group of patients, carbitocin 100 mcg will be given iv infusion over one minute after delivery of the head in cesarean section.
  Other Names: Carbetocin
  Arms: Pabal ( carbetocin)
Drug: Oxytocin 5 IU iv infusion and Methtergine 0.2 mg iv — In the second group of patients oxytocin 5 IU will be given iv infusion and Methergine 0.2 mg iv
  Other Names: Oxytocin and Methyl ergometrine
  Arms: Oxytocin and Methergine (methyl ergometrine)

SUMMARY:
The investigators compare the effectiveness and adverse effects of I.V carbetocin versus oxytocin & ergometrine I.V for prevention of postpartum haemorrhage following cesarean section.

DETAILED DESCRIPTION:
* Postpartum hemorrhage (PPH) accounts for nearly one quarter of all maternal deaths worldwide 1 and was the second most frequent cause of maternal death in the UK for the 2000-2002 triennium.
* Caesarean section is a recognized risk factor for PPH and the worldwide caesarean delivery rate is increasing .2
* A combination of oxytocin and ergometrine is effective in preventing postpartum hemorrhage but is frequently associated with side effects such as retained placenta and hypertension.
* A recent guideline on PPH prevention developed by the World Health Organization recommended the use of oxytocin for prevention of PPH in settings in which active management of labor is not practiced.
* Ergometrine is an ergot alkaloid and hypertension and cardiac disease are contraindications due to the possible development of severe hypertension and myocardial ischemia.
* Carbetocin is a newly developed uterotonics and it may represent a promising choice as reported in the literature. It is a synthetic analogue of human oxytocin with structural modifications that increase its half-life thereby prolonging its pharmacological effects .
* A prospective double blinded randomized study . The study population will include 200 patients. The study will take place in Beni_suef University Hospitals.
* Inclusion criteria:

  • Women with a singleton pregnancy undergoing elective caesarean section after 37 weeks of gestation.
* Exclusion criteria

  * Women undergoing cesarean section with general anesthesia will be excluded, because carbetocin is licensed for use with regional anaesthesia only.
  * women undergoing cesarean section at less than 37 weeks of gestation (likely to be emergency cesarean sections; a different smaller group from term pregnancies)
  * Hypertension with pregnancy.
  * Cardiac and coronary diseases with pregnancy
* Women included in the study were divided into 2 groups:

.Group (A): including 100 patients who will receive carbetocin 100 µg I.V after delivery of the fetal head.

.Group (B): including 100 patients who will receive a combination of intraoperative oxytocin 5 I.U & ergometrine 0.2 mg.

ELIGIBILITY:
Inclusion Criteria:

* • Women with a singleton pregnancy undergoing elective cesarean section after 37 weeks of gestation.

Exclusion Criteria:

* Women undergoing cesarean section with general anesthesia will be excluded, because carbetocin is licensed for use with regional anaesthesia only.
* women undergoing cesarean section at less than 37 weeks of gestation (likely to be emergency cesarean sections; a different smaller group from term pregnancies)
* Hypertension with pregnancy.
* Cardiac and coronary diseases with pregnancy

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Uterine tone and size | One hour after the cesarean section
  The uterine tone and size will be assessed by using a hand resting on the fundus and palpating the anterior wall of the uterus one hour after the operation. The presence of a boggy uterus with either heavy vaginal bleeding or increasing uterine size can suspect diagnosis of uterine atony.

SECONDARY OUTCOMES:
Blood loss | One hour after cesarean section
  Blood loss will be estimated postoperatively by giving each woman of each group standard 2 dressings (standard weight of dressing is 25 gm) for one hour postoperative and recording weight of blood soaked dressings and volume of lost blood.

OTHER OUTCOMES:
Hemoglobin concentration | Before and 24 hours after the operation
  Changes in hemoglobin concentrations before and 24 hours postoperative. Using a 10% fall in hematocrit value to define post-partum hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Nesreen Abdel Fattah Abdullah Shehata, Cairo, Egypt

REFERENCES:
- See also: Epidemiology of postpartum haemorrhage: a systematic review. Carroli G1, Cuesta C,2008 Dec;22(6):999-1012. doi: 10.1016/j.bpobgyn.2008.08.004. Epub 2008 Sep 25. Abalos E, Gulmezoglu AM. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Carroli+et+al.%2C+2008
- See also: • Villar J, Valladares E, Wojdyla D, Zavaleta N, Carroli G, Velazco A, et al. Caesarean delivery rates and pregnancy outcomes: the 2005 WHO global survey on maternal and perinatal health in Latin America. Lancet 2006; 367:1819-29. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Villar+JWojdylaC+Zavaleta+NC+Carroli+Velazco+Aetal.Cessarean+delivery+rates+and+pregnancy+outcomes%3A+the+2005+WHO+global+survey+on+maternal+and+perinatal+health+in+